CLINICAL TRIAL: NCT03677622
Title: Which Goal for Fluid Therapy During Colorectal Surgery is Followed by the Best Outcome: Near Maximal Stroke Volume or Restricted Fluid Therapy
Brief Title: Restrictive or Doppler-guided Fluid Treatment in Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holbaek Sygehus (Other)
Collaborators: Bispebjerg Hospital (Other); Glostrup University Hospital, Copenhagen (Other); Aarhus University Hospital (Other); Vejle Hospital (Other); Svendborg Hospital (Other)
Responsible Party: Principal Investigator, Birgitte Brandstrup, Sponsor, Holbaek Sygehus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Fluid Overload
Keywords: Restricted fluid therapy; Goal directed fluid therapy; Colorectal surgery; Surgery; Enhanced recovery; Fluid therapy
MeSH Terms: conditions — Edema

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stroke volume (SV) group (Experimental): As bellow but with the addition of HES (Voluven (R)) to near maximal stroke volume of the heart:
  A bolus injection of 200 ml Voluven® is given repeatedly with measurement of the SV until the increase in SV in response to the bolus is <10%.
  The Case Report File give detailed instructions for the interpretation of the SV during changes in position of the patient during laparoscopic surgery.
  Interventions: Drug: Voluven to near maximal stroke volume of the heart
- Restricted group (Active Comparator): Preoperatively: Clear oral fluids until 2 h before surgery. During surgery: If preoperative fluid intake <500 ml, NaCl 0.9% is given until 500 ml.
  Lost blood is replaced volume by volume with HES (Voluven®) with allowance of 500 ml extra.
  Postoperative fluid: The rest of the day of surgery, fluid is given to meet the basic needs, i.e. 1000 ml K-Na-glucose, K-glucose or glucose 5%. The patient is encouraged to drink and eat as soon possible.
  In the surgical department, fluid charts and weight changes monitor fluid balance. A body weight increase of two kilograms is allowed.
  Fluid losses is replaced with a fluid having a similar electrolyte composition as the loss and in an equal volume. If the weight increases more than two kilogram, furosemide is given to increase the diuresis.
  Interventions: Drug: Voluven to near maximal stroke volume of the heart

INTERVENTIONS:
Drug: Voluven to near maximal stroke volume of the heart — Stroke volume guided fluid treatment with Voluven on the basis of restricted fluid therapy

SUMMARY:
This is a clinical randomised double blinded multicentre trial of two different fluid treatments during colorectal surgery in an enhanced recovery programme A restricted fluid regimen aiming at zero fluid balance and less than two kilograms bodyweight change was compared with another fluid regimen where intravenous fluids were given to reach near maximal stroke volume of the heart, guided by a Doppler in the oesophagus.

The primary outcome was a composite outcome of postoperative complications and death.

Included was 150 patients undergoing elective colorectal surgery. No difference was found between the two groups. Both fluid therapies resulted in low complication rates. The difference in fluid volume between the groups was only 600 ml on the day of operation.

The results are published, see reference section.

DETAILED DESCRIPTION:
Background Hypovolemia can cause postoperative complications, circulatory collapse and death, regardless if the cause is blood loss or loss of other fluids. Therefore, doctors are giving fluid intravenously to patients undergoing surgery, and often in an amount larger than the measured losses. Recent studies, however, have shown that also fluid overload plays a part in complication development after surgery (1-3). It is therefore important to find the optimal fluid treatment for surgical patients.

In Denmark, approximately 3500 patients are undergoing surgery every year for colorectal cancer, and in addition, operations are performed for benign diseases. However, the complication rate after colorectal surgery remains high (approximately 30%).

Disagreement about which fluid treatment is optimal exist between three "schools for fluid therapy":

1. "Standard fluid therapy" which in addition to replacing external fluid loss (blood loss, urine and evaporation) include fluid to replace a "third space loss" and fluid to counteract low blood pressure (4-5). Standard therapy is poorly defined and differ between hospitals. It cause a bodyweight increase by 3-6 kilo (6-7).
2. "Goal-directed fluid therapy", where volume is given in a bolus injection of a colloid (typically hydroxyethyl starch (HES)) in order to keep the patient's stroke volume (SV) at a near maximum level (1). The heart is brought close to maximum performance. In theory, hypovolemia is prevented and oxygen supply to the tissues increased. In the studies available, HES is given on top of "standard therapy" and "Goal-directed fluid therapy" therefore result in a weight gain not measured in the available studies.
3. "Restrictive fluid therapy", replace only measurable fluid losses and strive to maintain the patient's normal (preoperative) body weight. The hypothesis is that excess fluid cause interstitial edema which may be harmful to the healing of tissue and function. (2,3,8).

   "Standard fluid therapy" is meaningful if a benefit exists in giving fluid to a possible third space loss and treat the vasodilatation caused by epidural analgesia by volume. However, a recent critical review of the literature poses serious doubts about the existence of a third space loss (9), and no beneficial effect of volume treatment of the vasodilatation caused by epidural analgesia been shown.

   "Goal-directed fluid therapy" tests the hypothesis that a near maximal stroke volume (SV) during surgery improves tissue oxygen supply, thus preventing the harmful effects of hypovolemia. Unfortunately, all studies that have tested "goal-directed fluid therapy" with esophageal Doppler monitoring have chosen to use a not well-defined "standard fluid regime" as their control group, and in the intervention groups they have chosen to first provide "standard fluid therapy" and then give a further HES to maximum stroke volume (10-16). In addition, length of hospital stay (LOS) were the primary endpoint not morbidity or mortality, and patients were not followed after discharge. The results of these studies differ. Most studies have shown shorter LOS in the intervention group, but only 3 of the studies have been blinded (11, 13, 16). Some studies have shown a lower complication rate in the intervention groups (12, 13, 16) some studies have not shown a difference in complication rate (10, 14, 15, 17) and some have raised suspicions that the intervention has been harmful, with increased mortality (15, 18).

   "Restrictive fluid treatment" is based on the following logic: If there is no third space loss, it is pointless to give saline to replace it, and if epidural vasodilatation is not corrected with volume, it is pointless to give fluid to increase BP.

   The hypothesis is that fluid overload might result in interstitial edema, harmful to tissue healing and cardiovascular function.

   Only a few studies have tested the effect of "restrictive fluid treatment" on the development of complications following major surgical procedures, but the results have been consistent: "Restrictive fluid treatment" has reduced the complication rate after elective abdominal surgery (2, 3).

   Purpose To investigate whether perioperative fluid therapy controlled by esophageal Doppler monitoring reduces postoperative complications compared to perioperative fluid therapy controlled by measuring external fluid loss and body weight.

   In addition, to investigate whether patients receiving "restrictive fluid therapy" develop hypovolemia with reduced SV during surgery.

   Design Clinical randomized double-blinded multicenter study, stratified for each center, and for laparoscopic and open surgery. This will result in a simultaneous stratification of combined epidural and general anesthesia (used in open surgery) and general anesthesia alone (as used in laparoscopic surgery).

   The patients are block randomized with a number of patients in each block unknown to the doctors performing the randomization. Several centers are participating to complete the trial within a reasonable time.

   The patients are following an enhanced recovery program in both arms.

   Material 150 patients undergoing elective colorectal resection will be included. The number was determined using data from complication databases, which shows a postoperative complication rate of approximately 30%. 2α is set at 5% and β is set at 15%, increasing the credibility of a possible negative result.

   A number of n > 67.5 patients in each group was calculated, and inclusion of 75 patients in each group (total 150 patients) was decided.

   Outcome The composite endpoint of mortality and postoperative complications is the primary endpoint.

   An event is accepted as a complication if it demands clinical treatment and fulfills given diagnostic criteria.

   Based on the following hypotheses; subgroup analysis are planned:

   Both hypovolemia and hypervolemia may be harmful to the cardiac function (low oxygen supply and congestion) and cause cardiovascular complications such as:

   • Newly developed arrhythmias, AMI, pneumonia, pulmonary congestion, newly developed pleural exudation, pulmonary edema or ARDS.

   Both hypovolemia and hypervolemia may be harmful to tissue healing (low oxygen supply and interstitial edema) and cause complications related to tissue healing and infection:

   • Infections of the wound, bursting of the wound (superficial and deep), leakage from the anastomosis and separation of a stoma.

   In addition, data for physiological changes in HR, BP, SV, Hemoglobin concentration, diuresis etc. will be analyzed.

   Method:

   A trial profile will account for all patients undergoing elective colorectal resections in the inclusion period. I.e. all patients undergoing elective colorectal resections must be consecutively screened for inclusion and asked to participate if no exclusion criteria is met.

   The information will take place the day before surgery. The information will be based on the written information (see appendix), and will be given in an easily understandable language and in an appropriate manner adapted to the individual.

   Patients are randomized to either "restrictive fluid treatment" (R group) or "fluid treatment to maximum SV" (SV group).

   Preoperative fluid treatment: All patients may drink until 2 hours before anesthesia. If supplemental intravenous fluids are needed, it is given in accordance with the loss, i.e.: Glucose isotonic (5%) replaces insensible perspiration (if diabetes insulin and if needed potassium is added). Registration of fluid intake begins at midnight on the day of the operation.

   Perioperative monitoring: Standard anesthesia monitoring as recommended by the Danish Anesthesiological Society is used. A catheter in the radial artery monitor the BP and is used for blood sampling. BP and HR are measured at least 3 times before induction of anesthesia and every five minutes during anesthesia.

   Immediately after the induction of anesthesia, all patients have a Doppler placed in the esophagus to measure the flow rate in the aorta, thereby calculating the stroke volume (SV). The SV is measured before surgery is started, and every 15 minutes throughout the operation.

   In the "Restrictive Group", the Doppler measurements are recorded to a black box (see later).

   Anesthesia: Routine premedication is given.

   In open surgery, combined epidural and general anesthesia are used:

   The Epidural catheter is inserted at the Th8-Th10 level, tested, and a continuous infusion of Bupivacaine 0.5% is running until sufficient blockade.

   General anesthesia is induced with Thiopental / Propofol, Fentanyl and Rocuronium (Esmerone®) for a neuromuscular blockade.

   Anesthesia is maintained with Sevoflurane / Fentanyl or Propofol / Remifentanil (Ultiva®).

   For laparoscopic surgery, only general anesthesia is used. In case of conversion from laparoscopic to open surgery, an epidural catheter is placed postoperatively.

   Perioperative fluid treatment: If the preoperative fluid intake <500 ml. it is supplemented to 500 ml. with saline in both groups. In addition, saline is given with the medicine.

   Lost blood is replaced volume by volume with HES (Voluven ®) with an allowance of 500 ml extra.

   In the SV group, a bolus injection of 200 ml Voluven® is given until the increase in SV is <10%.

   Blinding: Only the anesthesiologist know the randomization group and perioperative fluid treatment. It is unknown to the patient and to the project surgeon.

   As all patients in the study will receive NaCl 0.9%, Voluven ®, and other IV fluids, and as all patients are monitored with a Doppler in the esophagus, effective blinding of the surgeons can be achieved.

   In order to avoid bias of the anesthesiologist, the SV measurements are recorded to a black box in the restrictive group.

   Postoperative fluid treatment: Throughout the rest of the day of the operation, fluid is given to meet the basic needs, i.e. approx. 1000 ml K-Na-glucose, K-glucose or glucose 5%. The patient is encouraged to drink and eat as soon as it is safe to swallow.

   Nutrition is started as soon as possible (preferably in recovery) with protein drinks.

   In the surgical department, fluid charts and weight changes, allowing a body weight increase of two kilograms without treatment, monitor fluid treatment.

   If the weight increases more than two kilogram, furosemide is given to increase the diuresis.

   The patient's body weight is measured in the morning before surgery, and then every morning until discharge or the seventh post-operative day. The same set of scales are used throughout the course.

   Blood tests: Venous blood is taken in the morning on the day of the operation and every morning the following 5 days or until the patient is discharged.

   Surgery: Patients are operated with either open or laparoscopic technique. Antibiotic prophylaxis follows the department's routine. The bowel is not cleansed except for an enema before rectal surgery.

   Postoperative analgesia: In open surgical procedures, continuous, patient-controlled, epidural analgesia is given for a maximum of 4 days.

   In addition 1 g Paracetamol is given x 3-4, and / or Ibuprofen 400 mg x 3-4 if there are no contraindications. Supplemental Morphine p.n. is allowed.

   Nausea is treated with Ondansetron, Metoclopramide or DHB, depending on the cause of the patient's nausea. In case of suspicion of ventricular retention, a ventricular tube is applied for suction.

   Data collection The project doctor or surgeon see the patient every day and evaluates the patient's condition, prescribes fluid treatment, and assesses the presence and treatment of any complications.

   In addition, the patient is visiting the outpatient clinic approximately 30 days postoperatively. Any complications after discharge is recorded.

   Analysis

   The following analysis are planned:
   * "Intention-to-treat analysis" analyses all included patients for the primary endpoint.
   * "Per-protocol analysis" analyses those patients who have not been excluded following randomization (to be completed at > 10 exclusions only)
   * Analyzes of the above subgroups.
   * Analysis of the physiological data

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for colorectal resections if it is preoperatively estimated that the surgery may be cancer radical.
* ASA level 1-4.

Exclusion Criteria:

* Emergency surgery,
* Alcohol consumption > 5 units daily,
* Inability to give informed consent (language problems, unconscious, psychosis (including confusion))
* Pregnant and lactating women
* Contraindication for the use of HES (severe renal impairment, allergy, severe bleeding disorders and pregnancy)
* Other non-radically treated malignant diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2008-03-01 (Actual); Primary Completion 2009-07-31 (Actual); Study Completion 2009-08-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with a postoperative complication | 30 day follow-up
  Only complications demanding surgical or medical treatment. Diagnostic criteria for each complication was given by protocol

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte Brandstrup, PhD, Principal Investigator — Holbaek Sygehus

IPD SHARING:
Plan to Share IPD: Undecided
No plan

REFERENCES:
- [Background] Brandstrup B, Engquist A. [Is postoperative mortality affected by liberal intravenous fluid therapy? Presentation of a Cochrane analysis and a literature review]. Ugeskr Laeger. 2003 Mar 24;165(13):1342-5. No abstract available. Danish. PMID 12703278
- [Background] Brandstrup B, Tonnesen H, Beier-Holgersen R, Hjortso E, Ording H, Lindorff-Larsen K, Rasmussen MS, Lanng C, Wallin L, Iversen LH, Gramkow CS, Okholm M, Blemmer T, Svendsen PE, Rottensten HH, Thage B, Riis J, Jeppesen IS, Teilum D, Christensen AM, Graungaard B, Pott F; Danish Study Group on Perioperative Fluid Therapy. Effects of intravenous fluid restriction on postoperative complications: comparison of two perioperative fluid regimens: a randomized assessor-blinded multicenter trial. Ann Surg. 2003 Nov;238(5):641-8. doi: 10.1097/01.sla.0000094387.50865.23. PMID 14578723
- [Background] Nisanevich V, Felsenstein I, Almogy G, Weissman C, Einav S, Matot I. Effect of intraoperative fluid management on outcome after intraabdominal surgery. Anesthesiology. 2005 Jul;103(1):25-32. doi: 10.1097/00000542-200507000-00008. PMID 15983453
- [Background] Lobo DN, Stanga Z, Simpson JA, Anderson JA, Rowlands BJ, Allison SP. Dilution and redistribution effects of rapid 2-litre infusions of 0.9% (w/v) saline and 5% (w/v) dextrose on haematological parameters and serum biochemistry in normal subjects: a double-blind crossover study. Clin Sci (Lond). 2001 Aug;101(2):173-9. PMID 11473492
- [Background] Rasmussen LA, Rosenberg J, Crawford ME, Kehlet H. [Perioperative fluid therapy. A quality control study]. Ugeskr Laeger. 1996 Sep 16;158(38):5286-90. Danish. PMID 8966776
- [Background] Lobo DN, Bostock KA, Neal KR, Perkins AC, Rowlands BJ, Allison SP. Effect of salt and water balance on recovery of gastrointestinal function after elective colonic resection: a randomised controlled trial. Lancet. 2002 May 25;359(9320):1812-8. doi: 10.1016/S0140-6736(02)08711-1. PMID 12044376
- [Background] Brandstrup B, Svensen C, Engquist A. Hemorrhage and operation cause a contraction of the extracellular space needing replacement--evidence and implications? A systematic review. Surgery. 2006 Mar;139(3):419-32. doi: 10.1016/j.surg.2005.07.035. PMID 16546507
- [Background] Conway DH, Mayall R, Abdul-Latif MS, Gilligan S, Tackaberry C. Randomised controlled trial investigating the influence of intravenous fluid titration using oesophageal Doppler monitoring during bowel surgery. Anaesthesia. 2002 Sep;57(9):845-9. doi: 10.1046/j.1365-2044.2002.02708.x. PMID 12190747
- [Background] Gan TJ, Soppitt A, Maroof M, el-Moalem H, Robertson KM, Moretti E, Dwane P, Glass PS. Goal-directed intraoperative fluid administration reduces length of hospital stay after major surgery. Anesthesiology. 2002 Oct;97(4):820-6. doi: 10.1097/00000542-200210000-00012. PMID 12357146
- [Background] Mythen MG, Webb AR. Perioperative plasma volume expansion reduces the incidence of gut mucosal hypoperfusion during cardiac surgery. Arch Surg. 1995 Apr;130(4):423-9. doi: 10.1001/archsurg.1995.01430040085019. PMID 7535996
- [Background] Noblett SE, Snowden CP, Shenton BK, Horgan AF. Randomized clinical trial assessing the effect of Doppler-optimized fluid management on outcome after elective colorectal resection. Br J Surg. 2006 Sep;93(9):1069-76. doi: 10.1002/bjs.5454. PMID 16888706
- [Background] Sinclair S, James S, Singer M. Intraoperative intravascular volume optimisation and length of hospital stay after repair of proximal femoral fracture: randomised controlled trial. BMJ. 1997 Oct 11;315(7113):909-12. doi: 10.1136/bmj.315.7113.909. PMID 9361539
- [Background] Venn R, Steele A, Richardson P, Poloniecki J, Grounds M, Newman P. Randomized controlled trial to investigate influence of the fluid challenge on duration of hospital stay and perioperative morbidity in patients with hip fractures. Br J Anaesth. 2002 Jan;88(1):65-71. doi: 10.1093/bja/88.1.65. PMID 11881887
- [Background] Wakeling HG, McFall MR, Jenkins CS, Woods WG, Miles WF, Barclay GR, Fleming SC. Intraoperative oesophageal Doppler guided fluid management shortens postoperative hospital stay after major bowel surgery. Br J Anaesth. 2005 Nov;95(5):634-42. doi: 10.1093/bja/aei223. Epub 2005 Sep 9. PMID 16155038
- [Background] Price JD, Sear JW, Venn RM. Perioperative fluid volume optimization following proximal femoral fracture. Cochrane Database Syst Rev. 2004;(1):CD003004. doi: 10.1002/14651858.CD003004.pub2. PMID 14974001
- [Result] Brandstrup B, Svendsen PE, Rasmussen M, Belhage B, Rodt SA, Hansen B, Moller DR, Lundbech LB, Andersen N, Berg V, Thomassen N, Andersen ST, Simonsen L. Which goal for fluid therapy during colorectal surgery is followed by the best outcome: near-maximal stroke volume or zero fluid balance? Br J Anaesth. 2012 Aug;109(2):191-9. doi: 10.1093/bja/aes163. Epub 2012 Jun 17. PMID 22710266
- See also: Textbook, reference number 4 — http://bog.nu/titler/rationel-vaeske-elektrolytbehandling-og-ernaering-allan-engquist-og-birgitte-brandstrup
- See also: Textbook, reference number 5 — https://www.eu.elsevierhealth.com/millers-anesthesia-2-volume-set-9780443069598.html?gclid=EAIaIQobChMIiuLy6LnE3QIVFeh3Ch3i0wYeEAQYAiABEgInd_D_BwE